CLINICAL TRIAL: NCT03041285
Title: Phase I Study of Idronoxil Combined With Radiation Treatment in Men With Metastatic Prostate Cancer
Brief Title: Idronoxil Suppository Combine With Radiotherapy for Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: have difficulty finding eligible participants
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Thomas Eade, Principal Investigator, Royal North Shore Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOX66 version 1
Record Dates: First submitted 2017-01-20; First posted 2017-02-02 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Castrate- Resistant Prostate Cancer
MeSH Terms: interventions — phenoxodiol; Suppositories; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Group 1 (6 participants) will receive 400mg of Idronoxil (NOX66) daily in the form of one suppository. Group 2 (6 participants) will receive 800mg of Idronoxil daily (two suppositories). Group 2 will only commence once all group 1 participants have completed their treatment course and have experienced no toxicity greater than grade 2 according CTCAE version 4.03 for adverse events assessment.
Masking Description: There is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 NOX66 400mg and SBRT (Experimental): Group 1 patients will receive 400mg of Idronoxil (NOX66) suppository (1 suppository) daily from Day 0 (1 day before radiotherapy) until 7 days after completion of radiotherapy. Stereotactic Body Radiation Therapy will be given on Days1-5 (5 fractions). Total treatment course is 13-15 days, depends on whether radiotherapy is given on consecutive days or over the weekend.
  Interventions: Drug: idronoxil (NOX66) suppository; Radiation: Stereotactic Body Radiation Therapy
- Group 2 NOX66 800mg and SBRT (Experimental): Group 2 patients will receive 800mg of Idronoxil (NOX66) suppository (2 suppositories) daily from Day 0 (1 day before radiotherapy) until 7 days after completion of radiotherapy. Stereotactic Body Radiation Therapy will be given on Days1-5 (5 fractions). Total treatment course is 13-15 days, depends on whether radiotherapy is given on consecutive days or over the weekend.
  Interventions: Drug: idronoxil (NOX66) suppository; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: idronoxil (NOX66) suppository — Patients in Group 1 will be given 400mg of Idronoxil suppository (NOX66) (1 suppository) daily from Day 0(1 day before radiotherapy) until 7 days after radiotherapy. Group 2 will be given Idronoxil (NOX66) 800mg (2 suppositories) daily from Day 0 until 7 days after radiotherapy.
  All patients will receive one course of Stereotactic Body Radiation Therapy (SBRT), to be delivered in 20 Gray in 5 fractions.
  Radiotherapy session will involve irradiation of 1-2 lesions.
  .
  Other Names: NOX66
Radiation: Stereotactic Body Radiation Therapy — All patients (Group 1 and Group 2) will receive one course of Stereotactic Body Radiation Therapy (SBRT), to be delivered in 20 Gray in 5 daily fractions on consecutive days. Radiotherapy session (week 1) will involve irradiation to 1-2 lesions.

SUMMARY:
The aim of the study is to determine the toxicity of Idronoxil (NOX66) when used in combination with palliative radiotherapy for metastatic prostate cancer

DETAILED DESCRIPTION:
Who is it for? Patient may be eligible for this study if they have late stage metastatic prostate cancer which is castrate resistant and have metastatic lesions that are suitable for radiotherapy.

Study details There are two groups of patients in this study and no randomisation. The two groups will have two different doses of idronoxil (NOX66), representing a 2-step dose escalation. Both groups receive the same standard radiotherapy dose.

Group 1 will receive the lower dose (400 mg) of idronoxil suppository daily and Group 2 800 mg daily.

Recruitment into Group 2 will only commence once all Group 1 patients have completed the 13-day treatment course of idronoxil suppository without excessive unexpected toxicity. The total treatment duration will be 13-15 days for both groups depends on whether radiotherapy is given on consecutive days or over the weekend.

Day 0: commence idronoxil (NOX66) Days 1-5: 1 or 2 lesions will receive 20 Gy (radiotherapy dose unit) radiotherapy in 5 daily fractionated doses and continue daily NOX66 Day 6-12: Continue NOX66 (the duration of NOX66 will be 13-15 days depends on whether radiotherapy is given on consecutive days or over the weekend).

Both groups will have prostate-specific membrane antigen positron emission tomography (PSMA-PET) scans before starting treatment and three months after the last fraction of radiotherapy to assess treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed metastatic prostate cancer that is castrate-resistant.
* 2-3 lesions suitable for radiotherapy.
* ECOG Performance status 0-2.

  * Adequate bone marrow, hepatic and renal function
  * At least 4 weeks must have elapsed prior to commencement of idronoxil treatment since prior chemotherapy, investigational drug or biologic therapy

Exclusion Criteria:

* Chemotherapy regimens with delayed toxicity within the last 4 weeks.
* Any situation where the use of suppository therapy is contra-indicated or impractical(eg. chronic diarrhoea, colostomy, ulcerative colitis).
* No concurrent systemic chemotherapy or biologic therapy is allowed.
* Psychiatric disorder or social or geographic situation that would preclude study participation.
* Patient unable to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
safety of Idronoxil dose escalation | From start of NOX66 with stereotactic radiotherapy up to three months post treatment.
  Toxicity and relationship with study drug NOX66 will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) V4.3

SECONDARY OUTCOMES:
evidence of clinical tumour response | 3 months post treatment
  PSMA-PET CT will be done before and 3 months after treatment. The change in SUV in PSMA PET will be used to assess tumour metabolic response.
  Pre and post treatment tumour size on CT will be measured and RECIST criteria will be used to measure tumour response.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No